CLINICAL TRIAL: NCT01218646
Title: Safety and Immunogenicity Trial Among Adults Administered Quadrivalent Influenza Vaccine
Brief Title: Study of Quadrivalent Influenza Vaccine Among Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QIV03; UTN: U1111-1113-3619 (Other: WHO)
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-09

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent Inactivated Influenza Vaccine; Trivalent Inactivated Influenza Vaccine; Influenza viruses
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Investigational Quadrivalent Influenza Vaccine (Experimental): Participants will receive a dose of Investigational Quadrivalent Inactivated Influenza Vaccine
  Interventions: Biological: Investigational Quadrivalent Inactivated Influenza Vaccine, No Preservative
- Group 2: Investigational Trivalent Influenza Vaccine (Experimental): Participants will receive a dose of Investigational Trivalent Inactivated Influenza Vaccine
  Interventions: Biological: Investigational Trivalent Inactivated Influenza Vaccine, No Preservative
- Group 3: Licensed 2010-2011 Trivalent Influenza Vaccine (Active Comparator): Participants will receive a dose of Licensed 2010-2011 Trivalent Inactivated Influenza Vaccine
  Interventions: Biological: Fluzone®: 2010-2011 Trivalent Inactivated Influenza Vaccine, No Preservative
- Group 4: Licensed 2010-2011 Trivalent Influenza Vaccine (Active Comparator): Participants will receive a dose of Licensed 2010-2011 Trivalent Inactivated Influenza Vaccine
  Interventions: Biological: Fluzone®: 2010-2011 Trivalent Inactivated Influenza Vaccine, No Preservative

INTERVENTIONS:
Biological: Investigational Quadrivalent Inactivated Influenza Vaccine, No Preservative — 0.5 mL, Intramuscular
  Arms: Group 1: Investigational Quadrivalent Influenza Vaccine
Biological: Investigational Trivalent Inactivated Influenza Vaccine, No Preservative — 0.5 mL, Intramuscular
  Arms: Group 2: Investigational Trivalent Influenza Vaccine
Biological: Fluzone®: 2010-2011 Trivalent Inactivated Influenza Vaccine, No Preservative — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Group 3: Licensed 2010-2011 Trivalent Influenza Vaccine
Biological: Fluzone®: 2010-2011 Trivalent Inactivated Influenza Vaccine, No Preservative — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Group 4: Licensed 2010-2011 Trivalent Influenza Vaccine

SUMMARY:
The aim of the study is to evaluate a prototype quadrivalent influenza vaccine (QIV), the licensed 2010-2011 trivalent influenza vaccine (TIV) containing the primary B strain, and the investigational TIV containing the alternate B strain in adult subjects.

Primary Objective:

* To demonstrate non-inferiority of antibody responses to QIV compared with licensed 2010-2011 TIV (containing the primary B strain) and investigational TIV (containing the alternate B strain) as assessed by geometric mean titer (GMT) ratios for each of the four virus strains separately among subjects 65 years of age and older

Observational Objective:

* To describe the safety profiles of TIV among subjects 18 years of age and older and QIV in subjects 65 years and older, as assessed by solicited injection site and systemic adverse events (AEs) collected for 7 days post-vaccination, unsolicited adverse events collected from 21 days post-vaccination, and adverse events of special interest and serious adverse events (SAEs) collected from Visit 1 to Visit 2.

DETAILED DESCRIPTION:
All participants will receive a single dose of their assigned vaccine during Visit 1. They will be followed up for safety and immunogenicity through Day 21 post-vaccination (Visit 2)

ELIGIBILITY:
Inclusion criteria:

* Subject is 18 years of age or older on the day of inclusion.
* Informed consent form (ICF) has been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks post-vaccination.

Exclusion criteria:

* Known pregnancy, or a positive urine pregnancy test.
* Currently breastfeeding a child.
* History of serious adverse reaction to any influenza vaccine.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination.
* Planned receipt of any vaccine between Visit 1 and Visit 2.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first study vaccination or during the course of the study.
* Receipt of any influenza vaccine since 01 August 2010 (including 2009 H1N1 monovalent vaccine).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Thrombocytopenia, bleeding disorder, or receipt of anticoagulants contraindicating intramuscular vaccination.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barré Syndrome (GBS).
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Any chronic illness that, in the opinion of the Investigator, is not well controlled or that may interfere with trial conduct or completion or with assessment of adverse events.
* Known seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug use that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (12):
- United States (12):
  - Hoover, Alabama
  - South Miami, Florida
  - Springfield, Missouri
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - San Antonio, Texas

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 08 October through 01 December 2010 in 12 clinic centers in the US.
Pre-assignment Details: A total of 739 participants who met all the inclusion criteria and none of the exclusion criteria were enrolled, randomized and vaccinated in the study.
Groups:
- Group 1 (Investigational Quadrivalent Influenza Vaccine): Participants aged 65 years and older who received the Investigational Quadrivalent Influenza Vaccine
- Group 2 (Investigational Trivalent Influenza Vaccine): Participants aged 65 years and older who received the Investigational Trivalent Influenza Vaccine
- Group 3 (Licensed Trivalent Influenza Vaccine): Participants aged 65 years and older who received the Licensed 2010-2011 Trivalent Influenza Vaccine
- Group 4 (Licensed Trivalent Influenza Vaccine): Participants aged 18 to less than 65 years who received the Licensed 2010-2011 Trivalent Influenza Vaccine.
Period: Overall Study
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Started | 225 | 225 | 225 | 64
Completed | 224 | 225 | 223 | 63
Not Completed | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 3 (Licensed Trivalent Influenza Vaccine): Participants aged 65 years and older who received the received the Licensed 2010-2011 Trivalent Influenza Vaccine
- Total: Total of all reporting groups
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine) | Total
Number analyzed (Participants) | 225 | 225 | 225 | 64 | 739
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 64 | 64
  >=65 years | 225 | 225 | 225 | 0 | 675
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.4 (5.7) | 72.8 (5.6) | 72.8 (5.3) | 46.0 (11.6) | 70.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 121 | 126 | 27 | 403
  Male | 96 | 104 | 99 | 37 | 336
Region of Enrollment [Number; unit: Participants]
  United States | 225 | 225 | 225 | 64 | 739

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or With Trivalent Influenza Vaccines With Corresponding B Strain in Participants Aged 65 Years and Older.
Description: Immunogenicity outcomes were assessed in serum samples by hemagglutination inhibition (HAI) assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
Time Frame: Day 21 post-vaccination
Population: Geometric mean titers to the influenza vaccine B antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the B antigens, including results reported as less or greater than lower limit of quantitation (<LLOQ or >ULOQ).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 0
Titers
  B/Brisbane/60/2008 (220, 0, 219, 0) | 73.8 [63.9 to 85.3] | NA [NA to NA] — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group | 57.9 [50.6 to 66.4] |
  B/Florida/04/2006 (220, 221, 0, 0) | 61.1 [52.5 to 71.2] | 54.8 [47.5 to 63.3] | NA [NA to NA] — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group |

2. Other Pre Specified Outcome: Seroconversion Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or With Trivalent Influenza Vaccines (TIV) With Corresponding B Strains in Participants Aged 65 Years and Older.
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as < 10.
  Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
Time Frame: Day 21 post-vaccination
Population: Seroconversion with respect to influenza vaccine B strains (corresponding B strains) was determined in randomized and vaccinated adult participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 0
Participants
  B/Brisbane/60/2008 (220, 0, 219, 0) | 63 | NA — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group | 41 |
  B/Florida/04/2006 (220, 221, 0, 0) | 73 | 69 [0 to 0] | NA [0 to 0] — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group |

3. Primary Outcome: Geometric Mean Titers Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or After Trivalent Influenza Vaccines Without Corresponding B Strain in Participants Aged 65 Years and Older.
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
Time Frame: Day 21 post-vaccination
Population: Geometric Mean Titers to the influenza vaccine B strains (cross-reactive antibody) were determined in randomized and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 0
Titers
  B/Brisbane/60/2008 (220, 221, 0, 0) | 73.8 [63.9 to 85.3] | 42.2 [36.5 to 48.7] | NA [NA to NA] — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group |
  B/Florida/04/2006 (220, 0, 219, 0) | 61.1 [52.5 to 71.2] | NA [NA to NA] — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group | 28.5 [24.6 to 33.0] |

4. Other Pre Specified Outcome: Seroconversion Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or With Trivalent Influenza Vaccines Without Corresponding B Strain in Participants Aged 65 Years and Older.
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥ 1:10 and ≥ four-fold increase in post-vaccination titers.
Time Frame: Day 21 post-vaccination
Population: Seroconversion to influenza vaccine B Strains (cross-reactive antibody) was determined in randomized and vaccinated participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 0
Participants
  B/Brisbane/60/2008 (220, 221, 0, 0) | 63 | 19 | NA — B/Brisbane/60/2008 influenza virus antigen was not in the vaccine administered to this group. |
  B/Florida/04/2006 (220, 0, 219, 0) | 73 | NA [0 to 0] — B/Florida/04/2006 influenza virus antigen was not in the vaccine administered to this group. | 20 [0 to 0] |

5. Primary Outcome: Geometric Mean Titers Against the Influenza Virus Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines (TIV) in Participants Aged 18 Years or Older
Description: as for outcome 3
Time Frame: Day 0 and Day 21 post-vaccination
Population: Geometric Mean Titers to the influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 59
Titers
  A/H1N1, Pre-vaccination | 21.7 [17.9 to 26.3] | 21.1 [17.5 to 25.5] | 24.8 [20.4 to 30.1] | 26.7 [17.7 to 40.2]
  A/H1N1, Post-vaccination | 231 [188 to 283] | 271 [221 to 331] | 269 [221 to 328] | 728 [515 to 1030]
  A/H3N2, Pre-vaccination | 52.3 [42.1 to 65.0] | 42.3 [34.9 to 51.4] | 48.3 [40.0 to 58.4] | 33.0 [22.1 to 49.1]
  A/H3N2, Post vaccination | 501 [422 to 593] | 360 [302 to 429] | 291 [243 to 347] | 503 [361 to 701]
  B/Brisbane, Pre-vaccination | 27.1 [23.3 to 31.5] | 28.5 [24.2 to 33.6] | 29.0 [25.0 to 33.7] | 18.9 [14.0 to 25.4]
  B/Brisbane, Post-vaccination | 73.8 [63.9 to 85.3] | 42.2 [36.5 to 48.7] | 57.9 [50.6 to 66.4] | 97.7 [75.0 to 127]
  B/Florida, Pre-vaccination | 20.2 [17.5 to 23.3] | 19.7 [17.2 to 22.6] | 18.7 [16.4 to 21.3] | 19.5 [14.5 to 26.3]
  B/Florida, Post-vaccination | 61.1 [52.5 to 71.2] | 54.8 [47.5 to 63.3] | 28.5 [24.6 to 33.0] | 48.6 [35.5 to 66.4]

6. Other Pre Specified Outcome: Seroprotection Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or With Trivalent Influenza Vaccines in Participants Aged 18 Years or Older.
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroprotection was defined as a pre-vaccination and post-vaccination titer ≥ 1:40 (l/dil)
Time Frame: Day 21 post-vaccination
Population: Seroprotection to vaccine antigens were determined in randomized and vaccinated participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 59
Participants
  A/H1N1 Pre-vaccination | 70 | 70 [0 to 0] | 78 [0 to 0] | 27 [0 to 0]
  A/H1N1 Post-vaccination | 201 | 203 [0 to 0] | 200 [0 to 0] | 58 [0 to 0]
  A/H3N2 Pre-vaccination | 129 | 119 [0 to 0] | 131 [0 to 0] | 27 [0 to 0]
  A/H3N2 Post-vaccination | 220 | 212 [0 to 0] | 209 [0 to 0] | 57 [0 to 0]
  B/Brisbane Pre-vaccination | 101 | 108 [0 to 0] | 108 [25.0 to 33.7] | 21 [0 to 0]
  B/Brisbane Post-vaccination | 171 | 133 [0 to 0] | 157 [0 to 0] | 54 [0 to 0]
  B/Florida Pre-vaccination | 75 | 67 [0 to 0] | 68 [0 to 0] | 18 [0 to 0]
  B/Florida Post-vaccination | 161 | 149 [0 to 0] | 101 [0 to 0] | 38 [0 to 0]

7. Other Pre Specified Outcome: Seroconversion Against Influenza Virus Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or With Trivalent Influenza Vaccines in Participants Aged 18 Years and Older
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroconversion was defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
Time Frame: Day 21 post-vaccination
Population: Seroconversion to influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 220 | 221 | 219 | 59
Participants
  A/A1N1 | 145 | 161 [0 to 0] | 146 [0 to 0] | 46 [0 to 0]
  A/A3N2 | 152 | 139 [0 to 0] | 122 [0 to 0] | 50 [0 to 0]
  B/Brisbane/60/2008 | 63 | 19 [0 to 0] | 41 [0 to 0] | 27 [0 to 0]
  B/Florida/04/2006 | 73 | 69 [0 to 0] | 20 [0 to 0] | 18 [0 to 0]

8. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or With Trivalent Influenza Vaccines.
Description: Solicited injection site reactions: Pain, Erythema and Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
  Grade 3 Injection site reactions: Pain - Significant; prevents daily activity; Erythema and Swelling >100 mm.
  Grade 3 solicited systemic reactions: Fever (Temperature) ≥102.1°F; Headache, Malaise, and Myalgia - Significant; prevents daily activity.
Time Frame: Day 0 up to day 21 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all randomized and vaccinated participants, safety population.
Measure: Number; unit: Participants
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Number analyzed (Participants) | 225 | 225 | 225 | 64
Participants
  Injection site Pain (224, 225, 224, 63) | 73 | 52 [0 to 0] | 64 [0 to 0] | 31 [0 to 0]
  Grade 3 Injection site Pain (224, 225, 224, 63) | 2 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection site Erythema (224, 224, 224, 63) | 6 | 3 [0 to 0] | 3 [0 to 0] | 3 [0 to 0]
  Grade 3 Injection site Erythema (224, 224, 224, 63 | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling (224, 224, 224, 63) | 4 | 0 [0 to 0] | 3 [0 to 0] | 5 [0 to 0]
  Grade 3 Injection site Swelling (224, 224, 224, 63 | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Fever (224, 225, 223, 63) | 3 | 2 [0 to 0] | 0 [0 to 0] | 2 [0 to 0]
  Grade 3 Fever (224, 225, 223, 63) | 1 | 1 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Headache (224, 225, 224, 63) | 30 | 26 [0 to 0] | 26 [0 to 0] | 16 [0 to 0]
  Grade 3 Headache (224, 225, 224, 63) | 1 | 1 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Malaise (224, 225, 224, 63) | 24 | 26 [0 to 0] | 14 [0 to 0] | 16 [0 to 0]
  Grade Malaise (224, 225, 224, 63) | 1 | 2 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Myalgia (224, 225, 224, 63) | 41 | 32 [0 to 0] | 41 [0 to 0] | 22 [0 to 0]
  Grade 3 Myalgia (224, 225, 224, 63) | 1 | 1 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) upto 21 days post-vaccination
Arm/Group | Group 1 (Investigational Quadrivalent Influenza Vaccine) | Group 2 (Investigational Trivalent Influenza Vaccine) | Group 3 (Licensed Trivalent Influenza Vaccine) | Group 4 (Licensed Trivalent Influenza Vaccine)
Serious Adverse Events (participants affected / at risk) | 0/225 | 1/225 | 2/225 | 0/64
Other Adverse Events (participants affected / at risk) | 73/225 | 52/225 | 64/225 | 31/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Investigational Quadrivalent Influenza Vaccine) (N=225) | Group 2 (Investigational Trivalent Influenza Vaccine) (N=225) | Group 3 (Licensed Trivalent Influenza Vaccine) (N=225) | Group 4 (Licensed Trivalent Influenza Vaccine) (N=64)
Retina detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1 (Investigational Quadrivalent Influenza Vaccine) (N=225) | Group 2 (Investigational Trivalent Influenza Vaccine) (N=225) | Group 3 (Licensed Trivalent Influenza Vaccine) (N=225) | Group 4 (Licensed Trivalent Influenza Vaccine) (N=64)
Injection site pain (General disorders) | 73/224 (73) | 52 (52) | 64/224 (64) | 31/63 (31)
Injection site Swelling (General disorders) | 4/224 (4) | 0/224 (0) | 3/224 (3) | 5/63 (5)
Headache (Nervous system disorders) | 30/224 (30) | 26/224 (26) | 26 (26) | 16/63 (16)
Malaise (General disorders) | 24/224 (24) | 14/224 (14) | 26 (26) | 16/63 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 41/224 (41) | 32 (32) | 41/224 (41) | 22/63 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.